CLINICAL TRIAL: NCT06506838
Title: A Prospective, Open-Label, Single-Arm Clinical Study of Anlotinib Combined With Doxorubicin Monotherapy and Radiotherapy as Neoadjuvant Treatment for Soft Tissue Sarcoma
Brief Title: Anlotinib Combined With Doxorubicin and Radiotherapy as Neoadjuvant Treatment for Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnlotinibSTS
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Soft Tissue Sarcoma; Doxorubicin; Radiotherapy
Keywords: Soft Tissue Sarcoma; doxorubicin; Radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): For patients with the soft tissue sarcoma, the treatment regimen includes doxorubicin monotherapy with neoadjuvant and adjuvant chemotherapy cycles, alongside anlotinib and stereotactic body radiation therapy before surgery, followed by radical resection.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — For patients with the soft tissue sarcoma, the standard doxorubicin monotherapy regimen involves administering 37.5 mg/m² intravenously on days 1-2 of every 3 week . The treatment includes 3 cycles of neoadjuvant chemotherapy before surgery and 3 cycles of adjuvant chemotherapy after surgery, totaling 6 cycles. Anlotinib is administered at 12mg/d QD，day1~14, 21d/cycle. Neoadjuvant radiotherapy is conducted before surgery, starting after the second chemotherapy cycle, using stereotactic body radiation therapy (SBRT) with a dose of 4*10 Gy. Radical resection surgery is performed after the third chemotherapy cycle.

SUMMARY:
Exploring the Efficacy and Safety of Anlotinib Combined with Doxorubicin Monotherapy and Radiotherapy as Neoadjuvant Treatment for Soft Tissue Sarcoma

DETAILED DESCRIPTION:
This is a a prospective, open-Label, and single-arm clinical study. This study aims to evaluate the efficacy and safety of using anlotinib in combination with doxorubicin monotherapy and radiotherapy as a neoadjuvant treatment for soft tissue sarcoma. For patients with the soft tissue sarcoma, the standard doxorubicin monotherapy regimen involves administering 37.5 mg/m² intravenously on days 1-2 of each 3-week cycle. The treatment includes 3 cycles of neoadjuvant chemotherapy (pre-surgery) and 3 cycles of adjuvant chemotherapy (post-surgery), totaling 6 cycles. Anlotinib (ALC) is administered at 12mg/d QD，day1~14, 21d/cycle. Neoadjuvant radiotherapy is conducted before surgery, starting after the second chemotherapy cycle, using stereotactic body radiation therapy (SBRT) with a dose of 4*10 Gy. Radical resection surgery is performed in the ninth week, after the third chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. ECOG Performance Status score of 0-1.
3. Histologically or cytologically confirmed diagnosis of high-grade soft tissue sarcoma (G2-G3), classified as moderately sensitive or higher to chemotherapy (or determined suitable for radiotherapy and chemotherapy by the investigator). Typically includes histological types such as synovial sarcoma, vascular sarcoma, adult fibrosarcoma, intramuscular chondrosarcoma, leiomyosarcoma, liposarcoma, undifferentiated pleomorphic sarcoma, hepatic undifferentiated embryonic sarcoma, and unclassified soft tissue sarcomas.
4. Clinical confirmation of soft tissue sarcoma suitable for surgical resection after multidisciplinary assessment.
5. Presence of at least one measurable lesion according to RECIST v1.1 assessment criteria and suitable for ≥40 Gy/f radiotherapy (or determined suitable for radiotherapy by the investigator).
6. Laboratory and other examinations:Hematology: Absolute neutrophil count ≥1500/μL, platelet count ≥100,000/μL. Pulmonary function: No respiratory difficulty at rest, no reduced exercise tolerance, resting pulse oximetry >94% in room air.

   Renal function (creatinine clearance or radioisotope GFR ≥70 mL/min/1.73 m² or serum creatinine within normal limits according to age/gender). Liver function (total bilirubin ≤1.5 × ULN, AST or ALT <2.5 × ULN). Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%.
7. Signed informed consent and good compliance.
8. Reproductive-age women must use reliable contraception or have a negative pregnancy test (serum or urine) within 7 days before enrollment and agree to use appropriate contraception during the study and for 8 weeks after the last dose of investigational drug.

Exclusion Criteria:

1. Active autoimmune disease or history of autoimmune disease.
2. Receipt of any form of anti-tumor treatment within 4 weeks prior to enrollment, including radiotherapy, chemotherapy, molecular targeted therapy (such as angiogenesis inhibitors like sunitinib, sorafenib, imatinib, famitinib, regorafenib), and immunotherapy (eligible if last anti-tumor drug was stopped ≥5 half-lives before enrollment), or participation in another interventional clinical trial.
3. History of or current simultaneous malignancy within 3 years, excluding cured lung cancer, cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumors), Tis (carcinoma in situ), and T1 (tumor invades lamina propria)].
4. Unresectable sarcomas, including severe vascular, neural, or bone involvement, or cases where complete surgical resection is not safely feasible.
5. Factors affecting oral medication (such as dysphagia, severe chronic diarrhea, and intestinal obstruction, etc.).
6. History of bleeding, with any grade 3 or higher bleeding event as per CTCAE 4.0 within 4 weeks before screening.
7. Uncontrolled diseases or past medical history, such as:

   * NYHA Class ≥2 heart failure, unstable angina, myocardial infarction within the past 12 months.
   * Active infections requiring systemic treatment.
   * Known HIV infection, syphilis history, psychiatric disorders (such as epilepsy and dementia), or substance abuse disorders.
   * Thromboembolic events (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism within the past 6 months before enrollment.
8. According to NYHA standards, Class III-IV heart failure, or left ventricular ejection fraction (LVEF) <50% on echocardiography.
9. Major surgery within 4 weeks prior to randomization or severe traumatic injury, fracture, or ulcer.
10. Long-standing unhealed wounds or fractures.
11. Pregnancy or lactation in women.
12. Known allergy to any investigational drug.
13. Investigator judgment that the subject has other factors that may lead to premature termination of the study, such as severe laboratory abnormalities, family or social factors affecting subject safety, or data and sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response rate | 3 months
  Typically defined as residual tumor cells ≤10% in the surgical specimen after treatment
Pathologic Complete Response rate | 3 months
  Absence of any residual tumor cells in the surgical specimen following treatment.

SECONDARY OUTCOMES:
Objective Response Rate | 3 months
  The proportion of patients in a clinical trial whose tumor size decreases (partial response) or disappears (complete response) after treatment.
Disease-Free Survival | 2 years
  The length of time during and after treatment that a patient lives with the disease without it progressing

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangdong provincial people's hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.